CLINICAL TRIAL: NCT00900835
Title: Reducing Barriers to Pain and Fatigue Management
Brief Title: Pain and Fatigue Management in Patients With Breast Cancer, Prostate Cancer, Colon Cancer, or Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Betty Ferrell, City of Hope Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 04140; R01CA115323 (NIH); P30CA033572 (NIH); CHNMC-04140; CDR0000628799 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Breast Cancer; Colorectal Cancer; Fatigue; Lung Cancer; Pain; Prostate Cancer
Keywords: fatigue; pain; recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent prostate cancer; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent colon cancer; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; extensive stage small cell lung cancer; limited stage small cell lung cancer; recurrent non-small cell lung cancer; recurrent small cell lung cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Fatigue; Lung Neoplasms; Pain; Prostatic Neoplasms; Colonic Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Early Intervention, Educational; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: educational intervention
Other: questionnaire administration
Other: study of socioeconomic and demographic variables
Procedure: assessment of therapy complications
Procedure: fatigue assessment and management
Procedure: quality-of-life assessment
Procedure: standard follow-up care

SUMMARY:
RATIONALE: Collecting information over time about patients' and health care providers' understanding of pain and fatigue and providing education about pain and fatigue management may improve quality of life.

PURPOSE: This clinical trial is studying pain and fatigue management in patients with breast cancer, prostate cancer, colon cancer, or lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To test the effects of the Passport to Comfort (Passport) intervention at 1 and 3 months post-intervention by comparing baseline data to the high-intensity intervention.
* To test the effects of select demographic and disease/treatment variables on outcomes of the Passport model at 1 and 3 months post-intervention compared to pre-intervention.
* To examine perceived patient and professional satisfaction with the Passport model.
* To test the effects of the Passport intervention by comparing high-intensity to low-intensity.

OUTLINE: Patients are stratified according to cancer diagnosis (breast vs prostate vs colon vs lung), pain level (< 4 vs ≥ 4 on pain scale), and fatigue level (< 4 vs ≥ 4 on fatigue scale). Patients are assigned to 1 of 3 groups.

* Group 1 (enrolled during months 1-8): Patients undergo pain and fatigue assessment periodically by demographic and treatment data, Quality of life-Patient Tool, BQII, Piper Fatigue Scale, Pain and Fatigue Knowledge Tools, and Patient Satisfaction Tool. Patients receive usual care and undergo pain and fatigue evaluation with no algorithms or formal education. Research nurses conduct chart audits to identify professional and system barriers but receive no medical education, peer review, or feedback. Medical professionals undergo assessment periodically by a Demographic Data Tool, Pain and Fatigue Knowledge Tools, Chart Audit Tool, and Provider Satisfaction.
* Group 2 (enrolled during months 9-30): Patients and medical professionals are assessed periodically as in group 1. Patients undergo a high-intensity Passport intervention with algorithms based on National Comprehensive Cancer Network (NCCN) guidelines, pain and fatigue education once weekly for 4 weeks, and follow-up reinforcement phone calls every 2 weeks. Research nurses conduct chart audits of congruence between practice and guidelines, tape education sessions, and receive feedback from the principal investigator in the form of a Tape-Monitoring Checklist. Medical oncologists attend training on the use of the algorithms, peer review pain and fatigue management audit with feedback, and reinforce and apply content in clinical rounds.
* Group 3 (enrolled during months 34-57): Patients and medical professionals are assessed periodically as in group 1. Patients undergo a low-intensity Passport intervention as in group 2. Medical professionals conduct realistic implementation of the intervention into existing systems and procedures within the cancer center, less direct education and system intervention, and share group 2 experiences.

After completion of study intervention, patients are followed at 1 and 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast, prostate, colon, or lung cancer (any stage)

  * Diagnosed ≥ 1 month before study entry
* Reports pain and/or fatigue intensity ≥ 4 on a scale of 0-10
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Life expectancy ≥ 6 months
* Able to read and understand English

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2005-06; Primary Completion 2009-09 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Quality of life
Pain knowledge of patients and professionals
Fatigue knowledge of patients and professionals
Adherence to algorithm by patients, professionals, and system
Satisfaction of patients and professionals

CONTACTS AND LOCATIONS:
Overall Officials: Betty Ferrell, PhD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States